CLINICAL TRIAL: NCT05129163
Title: Associations Between Various Geriatric Syndromes and Nutrition Status and Dietary Pattern in Elderly
Brief Title: Effects of Community-center Based Dietary Intervention on Frailty Prevention and Regression in the Elderly.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the impacts of COVID-19, the study had to terminate.
Sponsor: Academia Sinica, Taiwan (Other)
Responsible Party: Principal Investigator, Wen-Harn Pan, Distinguished Research Fellow, Academia Sinica, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AS-IRB01-16057
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Placebo Comparator): The control group received weekly one-hour group exercise training for 3 months.
  Interventions: Behavioral: Exercise
- Exercise and nutrition (Experimental): The intervention group had weekly one-hour group exercise training the same as the control and an additional weekly one-hour group nutrition session for 3 months.
  Interventions: Behavioral: Exercise; Behavioral: Nutrition activities

INTERVENTIONS:
Behavioral: Exercise — The group exercise training was held in each community center. The group exercise training contained aerobic exercise, complex physical fitness exercise, muscle training, and balance and coordination training.
Behavioral: Nutrition activities — The intervention programs included: (a) training on-site staffs to use motivational interview techniques to communicate, to estimate participant's energy requirements, and to learn how to provide proper amounts of foods to individual elderlies, (b) nutrition grouped activities on ①know my plate, ②wholegrains, ③ drinking teas with dairy, and nuts, ④novel ways to eat fruit and vegetables, ⑤healthy breakfast ideas. In the first month, participants were intervened with the activities laid out above; in the second month, participants were intervened with qualitative discussion on elders' dietary changes; in the third month, participants were intervened with designed activities that helped break down barriers in order to establish a long-term change in dietary habits.
  Arms: Exercise and nutrition

SUMMARY:
Recent interventional studies have shown that frailty can be improved by modifying dietary quality. In this study, a set of nutrition-centric health promotion activities was developed in accordance with the Taiwanese Daily Food Guide for elderly participants of the community centers to improve their nutrition in everyday practice and examined the efficacy of these activities on slowing down the development or regression of frailty. The study was a cluster-randomized controlled trial. Recruited community centers were randomly assigned into either the control or the intervention group. The intervention period lasted for 3 months. Both the control and intervention groups received weekly one-hour group exercise training. The intervention group had an additional weekly one-hour group nutrition session. The intervention programs included: (a) training on-site staffs to use motivational interview techniques to communicate, to estimate participant's energy requirements, and to learn how to provide proper amounts of foods to individual elderlies, (b) nutrition grouped activities on ①know my plate, ②wholegrains, ③drinking teas with dairy, and nuts, ④novel ways to eat fruit and vegetables, ⑤healthy breakfast ideas. In the first month, participants were intervened with the activities laid out above; in the second month, participants were intervened with qualitative discussions on dietary changes; in the third month, participants were intervened with designed activities that helped break down barriers in order to establish a long-term change in dietary habits. Improvement in nutritional status was the primary outcome. Secondary outcomes included frailty scores, physical performance, and mental health. The measurements were performed at baseline, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Able to walk independently for 14 meters within 1 minute
* Willing to sign the informed consent

Exclusion Criteria:

* Under dietary control by doctors' instructions
* With mental illness, mental disorders, or unable to communicate
* With severe diseases such as under treatments for cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 219 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in intake frequency (portion per day) on the six food groups at months 3 and 6. | Baseline, Month 3 and Month 6
  The six food groups include:
  1. Whole grains and starchy vegetables
  2. Protein foods: soy beans, fish, eggs, and meat
  3. Vegetables
  4. Fruits
  5. Dairy
  6. Oils, nuts and seeds
Change from baseline in the ratios of concentration on urinary nutritional biomarkers at months 3 and 6. | Baseline, Month 3 and Month 6
  The concentrations of the following urinary nutritional biomarkers were determined: urinary urea nitrogen (mg/dL), urinary calcium (mg/dl), urinary potassium (mmol/L), urinary magnesium (mg/dL), and urinary creatinine (mg/dL).
  The urinary urea nitrogen to creatinine ratios, urinary calcium to creatinine ratios, urinary potassium to creatinine ratios, and urinary magnesium to creatinine ratios was estimated at baseline, moths 3 and 6.
Change from baseline in frailty status at months 3 and 6. | Baseline, Month 3 and Month 6
  Frailty status was defined using modified Linda Fried criteria with cutoff points from the investigators' previous intervention studies.
  Five frail phenotypes were assigned: (1) unintentional weight loss, (2) self-reported exhaustion, (3) weak grip strength, (4) slow gait speed, and (5) low level of physical activity. To estimate frailty, participants scored 1 point from each phenotype if any of these were satisfied; a maximum score of five was possible. Participants were classified by their point scores as follows: 'robust' for 0 point; 'pre-frail' for 1 or 2 points; and 'frail' for ≥3.

SECONDARY OUTCOMES:
Change from baseline in the score of digit span at months 3 and 6. | Baseline, Month 3 and Month 6
  A digit span task is used to measure working memory's number storage capacity. Subjects are read a sequence of numbers and asked to repeat the same sequence back to the examiner in order (forward span) or in reverse order (backward span). The score is the length of the longest correctly repeated sequence. The maximum number of digits in a sequence is 9 and the minimum number of digits in a sequence is 2. The higher scores mean a better outcome.
Change from baseline in the scores on the Geriatric Depression Scale at months 3 and 6. | Baseline, Month 3 and Month 6
  The Geriatric Depression Scale (GDS) is a self-report measure of depression in older adults. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, PhD, Principal Investigator — Academia Sinica, Taiwan
Locations (1):
- Institute of Biomedical Sciences, Academia Sinica, Taipei, Taiwan

REFERENCES:
- [Background] Hsieh TJ, Su SC, Chen CW, Kang YW, Hu MH, Hsu LL, Wu SY, Chen L, Chang HY, Chuang SY, Pan WH, Hsu CC. Individualized home-based exercise and nutrition interventions improve frailty in older adults: a randomized controlled trial. Int J Behav Nutr Phys Act. 2019 Dec 2;16(1):119. doi: 10.1186/s12966-019-0855-9. PMID 31791364
- [Background] Wu SY, Hsu LL, Hsu CC, Hsieh TJ, Su SC, Peng YW, Guo TM, Kang YW, Pan WH. Dietary education with customised dishware and food supplements can reduce frailty and improve mental well-being in elderly people: A single-blind randomized controlled study. Asia Pac J Clin Nutr. 2018;27(5):1018-1030. doi: 10.6133/apjcn.032018.02. PMID 30272850